CLINICAL TRIAL: NCT00281177
Title: Center for Reducing Asthma Disparities - Northwestern University/Cook County Hospital Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Purpose: Treatment
Other Study IDs: 1199; U01HL072478 (NIH); U01HL072496 (NIH)
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2006-06

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

INTERVENTIONS:
Behavioral: Asthma Disparity Reduction Strategy

SUMMARY:
The purpose of this study is to characterize the relationship of social stress, coping, and self-regulatory health behaviors in the context of asthma disparities among African American and low income populations.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a serious chronic condition affecting over 14 million Americans, but the prevalence rates are higher in certain populations (e.g. 10% in inner-cities and 30% among the homeless versus 5% in a general population of whites). African Americans and Hispanics from the Northeast are twice as likely to die from asthma as whites. African Americans are four times as likely to be hospitalized for asthma and are five times more likely than whites to seek care for asthma at an emergency department. Reasons for these higher rates are not certain, and most likely result from an interaction of risk factors, such as environmental exposures, genetic predisposition, access to appropriate medical care, socioeconomic status, and cultural health practices. The National Heart, Lung, and Blood Institute supports a variety of activities to address the pressing public health problems posed by asthma. However, progress in reducing disparities has been disappointingly slow. Separate, independent research projects have generated important clues for understanding the nature and scope of the problem. A more coordinated, interdisciplinary and comprehensive approach to research is needed to take advantage of these clues, move the science further and faster, and increase our capacity to improve health outcomes among minority and economically disadvantaged populations. Cooperative centers of research that foster partnerships among minority medical centers, research intensive institutions, and the communities in which asthma patients live will promote such advancement.

The Request for Applications for the Centers for Reducing Asthma Disparities was released in October 2001. The objective of the program is to promote partnerships (called centers) between a minority serving institution (MSI) that may not have a strong research program and a research intensive institution (RII) that has a track record of NIH-supported research and patient care. The purpose of the partnership is to conduct collaborative research on asthma disparities (i.e., greater prevalence of asthma, higher rates of morbidity due to asthma, and lesser access or use of quality medical care among minorities and poor).

DESIGN NARRATIVE:

The project will develop a collaborative research program between Northwestern University Feinberg School of Medicine and Cook County Hospital to fully characterize the relationship of social stress, coping, and self-regulatory health behaviors in the context of asthma disparities among African American and low income populations. Once characterized, the project will then develop and test an intervention strategy to reduce asthma disparities in high-risk populations based on evidence-based models that have demonstrated success in social work, nursing, and community interventions.

There are four research aims for the center: (1) To develop and validate culturally appropriate psychosocial instruments related to the underlying causes of disparity in asthma morbidity; (2) To identify the structural relationships of psychosocial factors to other known influential factors related to disparities in asthma outcomes; (3) To study the changes in structural relationship among influential factors in asthma disparity over time, as related to changes in health status; (4) To develop, pilot test, and field test a community-based asthma team (peer coach, asthma nurse, and social worker) intervention to enhance individuals ability to cope with chronic illness and improve asthma-related behaviors. A second major goal of the Center will be to train and mentor new clinical investigators and social scientists to be able to conduct research in this field of interest.

The study completion date listed in this record was obtained from the "Project End Date" entered in the Query View Report (QRV) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-09; Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Shannon, Principal Investigator — Hektoen Institute/Cook County Hospital; Kevin Weiss, Principal Investigator — Northwestern University Feinberg School of Medicine